CLINICAL TRIAL: NCT01755663
Title: Comparison of Efficacy and Safety of Ivabradine Versus Metoprolol for Controlling Heart Rate Prior to 640-Slice Computed Tomographic Angiography in Elective Patients
Brief Title: Comparison of Efficacy of Ivabradine Versus Metoprolol
Acronym: IMAGE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Col. Suthee Panichkul (Other)
Collaborators: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor-Investigator, Col. Suthee Panichkul, Col. Suthee Panichkul, Phramongkutklao College of Medicine and Hospital
Organization: Phramongkutklao College of Medicine and Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pharmongkutklao
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Artery Disease
Keywords: CT coronary; Coronary arterial disease; ivabradine; metoprolol
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ivabradine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Experimental): Patients will recieved ivabradine(5) 1 tab bid pc for 3 day and the day of CT, and recieve placebo of metoprolol
  Interventions: Drug: Ivabradine and Metoprolol
- metoprolol (Active Comparator): Metoprolol (100) 1/2 tab bid pc for 3 day and the day of CT coronary , and placebo of ivabradine
  Interventions: Drug: Ivabradine and Metoprolol

INTERVENTIONS:
Drug: Ivabradine and Metoprolol

SUMMARY:
Ivabradine may be better than Metoprolol for controlling heart rate before Coronary CTA.

ELIGIBILITY:
Inclusion Criteria:

* elective patient on scheduled for 640 slices CT coronary at Phramonkutklao hospital
* Resting heart rate > 70 BPM
* age > 18 years and informed consent

Exclusion Criteria:

* Heart rate > 100 BPM
* BP <100/60 mmHg
* recent congestive heart failure in 1 mo.
* SA node, AV node disease and AF
* on permanent pacemaker
* CrCL < 15ml/min. , AST or ALT > 3x UNL
* on HR reducing drug such as diltiazem, verapamil, digitalis
* contraindication for ivabradine or metoprolol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate of patient before CT coronary | 1 January 2013 to 31 december 2013

SECONDARY OUTCOMES:
safety and side effect of Metoprolol and Ivabradine | 1 january 2013 to 31 december 2013

OTHER OUTCOMES:
Image quality | 1 january 2013 to 31 december 2013

CONTACTS AND LOCATIONS:
Overall Officials: Purich - Surunchupakorn, M.D., Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramonkutklao Hospital, Bangkok, Thailand